CLINICAL TRIAL: NCT06988111
Title: A Prospective, Randomized Controlled Trial Comparing Noninvasive Ventilation (NIV) Versus High-Velocity Nasal Cannula (HVNC) in the Management of Acute Post-Operative Respiratory Failure
Brief Title: Management of Post-operative Respiratory Failure by Using NIV and High Velocity Nasal Insufflation (HVNI)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Shaddad, Associate Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 375690
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Failure Without Hypercapnia; Respiratory Failure With Hypercapnia; Postoperative Respiratory Complication
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: The patient with operative respiratory failure will be compared using NIV and High velocity nasal cannula devices
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-invasive Ventilation group (Experimental): NIV Arm
  * Device: Bi-level positive airway pressure (BiPAP) via oronasal mask.
  * Initial settings: inspiratory positive airway pressure (IPAP) 10 cmH₂O, expiratory positive airway pressure (EPAP) 5 cmH₂O, and fraction of inspired oxygen (FiO₂) titrated to oxygen saturation (SpO₂) ≥ 92%.
  * Weaning: Decrement IPAP/EPAP by 2 cmH₂O every four hours as tolerated.
  Interventions: Device: BIPAP
- High Velocity Nasal Cannula (HVNC) group (Experimental): HVNC Arm
  * Device: Heated, humidified high-flow nasal cannula (HFNC) system.
  * Initial flow: 50 L/min, fraction of inspired oxygen (FiO₂) titrated to SpO₂ ≥ 92%.
  * Weaning: Reduce flow by 10 L/min every 4 h as tolerated.
  Interventions: Device: Vapotherm

INTERVENTIONS:
Device: BIPAP — The second arm (NIV group) will be managed by BIPAP device for post-operative respiratory failure
  Arms: Non-invasive Ventilation group
Device: Vapotherm — The first arm (HVNC group) will be managed by Vapotherm device for post-operative respiratory failure
  Other Names: High-velocity nasal insufflation; High velocity nasal cannula
  Arms: High Velocity Nasal Cannula (HVNC) group

SUMMARY:
Postoperative respiratory failure (PORF) remains a critical driver of morbidity, mortality, and incremental care costs in surgical populations. Traditional escalation often involves invasive mechanical ventilation, which is associated with ventilator-associated pneumonia (VAP), prolonged intensive care unit (ICU) stays, and increased resource burden.

DETAILED DESCRIPTION:
Noninvasive ventilation (NIV) and high-flow nasal cannula (HFNC) have both been shown to improve oxygen levels effectively and reduce the need for reintubation in various patient groups. However, head-to-head data in patients with obstructive or restrictive pulmonary function (PORF) are scarce.

This protocol employs a robust and scalable design to generate high-quality evidence, empower perioperative stakeholders, and optimize patient-centric respiratory strategies. We hypothesize that NIV will reduce 72-hour reintubation rates compared to HFNC, translating into shorter ICU stays and lower costs.

Methodology & Operational Workflow

* Screening & Consent Identify eligible patients in the post-anesthesia care unit (PACU) or ICU. Obtain informed consent from the patient or legal surrogate.
* Baseline Assessment The baseline assessment includes demographics, comorbidities, and surgical data, as well as baseline arterial blood gases (ABG), vital signs, and comfort scores.
* Randomization & Initiation Allocate via a secure web-based randomization module. Initiate assigned respiratory support within 30 minutes of notification.
* Monitoring & Data Collection The patient is receiving continuous pulse oximetry and respiratory rate monitoring.

ABGs and fraction of inspired oxygen (FIO2) at 1 hour, 6 hours, and 24 hours. Comfort scores every six hours. Record interface-related adverse events.

- Escalation Criteria The patient exhibits persistent partial arterial oxygen pressure/fraction of inspired oxygen ratio (PaO2/FiO2) levels of less than 100, even at maximal settings.

Hemodynamic instability occurs due to the use of new-onset vasopressors. Deterioration leading to invasive ventilation → classified as "reintubation."

* Weaning Protocol. Transition to standard oxygen therapy when the flow or pressure is minimal.
* Follow-Up & Discharge Track ICU length of stay (LOS), hospital LOS, and ventilation-free days (VFD). Keep a record of the 30-day survival rate and any readmissions.
* Statistical Analysis Plan Primary Endpoint: Compare reintubation rates using a χ² test; report the risk difference and 95% confidence interval.
* Missing Data: Multiple imputation for datasets with ≤ 5% missing data; sensitivity analysis for worst-case scenarios.
* Interim Analysis: After 50% enrollment, the Data Safety and Monitoring Board (DSMB) reviews efficacy and futility, using O'Brien-Fleming boundaries.

ELIGIBILITY:
Inclusion criteria:

* Age above 18 years
* within 48 hours after major surgery
* PAO2/FIO2 less than 200
* Signs of respiratory distress and respiratory rate (RR) more than 25 cycles/minute

Exclusion Criteria:

* Age below 18 years
* Pregnant ladies
* Orofacial trauma or burns
* Active Gastrointestinal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Weaning success | At 48 hours and then daily for 28 days.
  The primary outcome will be comparing the weaning success (in days) for both arms of the study group. This will be accessed after 48 hours and on a daily basis until the weaning criteria are met or for 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M. Shaddad, MD, Principal Investigator — Assuit Univeristy; Aliae A. Hussien, MD, Principal Investigator — Assiut University
Locations (1):
- Assuit Univeristy, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data supporting the primary and secondary outcomes, along with accompanying data dictionaries and the statistical analysis plan, will be made available by Assiut University's institutional data-sharing policies.
Supporting Information: Study Protocol, SAP
Time Frame: 6-36 months after publication.
Access Criteria: Data will be accessible 6-36 months after publication to qualified researchers upon submission of a study proposal, approval by the University Research Ethics Committee, and execution of a data-use agreement.